CLINICAL TRIAL: NCT00367354
Title: Respiratory Motion Analysis in Children for Improvement of MR (Magnetic Resonance) Imaging of Congenital Heart Disease
Brief Title: Respiratory Motion Analysis in Children With MRI
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Other Study IDs: IRB00041134
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Congenital Disorders
Keywords: Imaging Technology; Cardiology
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to analyze the respiratory motion process as relevant in cardiac MRI imaging and apply the results for development of improved imaging methods and software correction. To accomplish this, we will develop an imaging protocol for monitoring respiratory motion.

The imaging protocol will be limited to less than five minutes of acquisition time so it may be performed as "piggyback" acquisition following clinically prescribed imaging studies on pediatric and adult cardiac MRI patients, but will also be applied to normal healthy volunteers.

Hypothesis Characterization of respiratory motion will help improve image quality by allowing optimized scan acquisition and retrospective correction of acquired data.

DETAILED DESCRIPTION:
Cardiac magnetic resonance imaging (MRI) is used heavily in the research setting but its use is limited in clinical practice, the main reason being artifact (noise) from respiratory and cardiac motion. To counteract these sources of motion, many different applications have been applied. For cardiac motion, ECG (electrocardiogram) gating is widely used, while respiratory motion reduction uses methods of breath holding or respiratory gating techniques.

Patients will be recruited based on whether they are a normal healthy volunteer or a patient already receiving a routine cardiac MRI.

Normal Healthy Volunteers Patients will be recruited via a flyer posted in various locations at Emory University. The contents of this flyer will adhere strictly to Emory IRB Advertisement guidelines. Subjects will register by contacting Marijn Brunner, PhD, by email or telephone.

Patients already scheduled for a routine cardiac MRI The MRI technical specialist will review the laboratory schedule daily. Those who are already scheduled for a routine cardiac MRI will be approached by a study staff member in the Children's MRI Department. The patient will be asked if he/she would wish to enroll in this study. The patient will be requested to sign a consent prior to any study procedures being performed.

MRI image data will be collected by the prescribed protocol for respiratory monitoring. All MRI data will be acquired by standard FDA approved imaging methods. The image data will be transferred by network to the Pediatrics Imaging Research Laboratory where they will be stored on a password-protected computer and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit two groups of patients - 35 healthy volunteers (21 years or older) and 25 cardiac MRI patients of different age groups.

We wish to recruit cardiac patients from Children's Healthcare of Atlanta into five (5) different categories defined by the overall characteristics of breathing motion. The categories are:

1. neonates/infants (shallow belly breathing)
2. young children (unable to do controlled breathing or breath-holding on command, up to approximately 7 years of age)
3. older children capable of controlled breathing/breath-holding on command (approximately 8-12 years of age)
4. teenagers/adolescents/young adults (ages 13 through 17)
5. adults (18 and older) These categories may be adjusted or modified during the project as deemed appropriate based on the analysis results.

We will recruit 10 - 35 healthy volunteer subjects for scans to define the MRI imaging protocol for respiratory motion monitoring. Healthy subjects are defined as those individuals who do not have a prior history of heart or lung disease nor are currently diagnosed with heart or lung disease. This information will be obtained verbally during the subject screening process.

Exclusion Criteria:

* No exclusion criteria will be placed on any sub-population based on age, gender or race other than the patient not freely giving written informed consent or having a history or current diagnosis of heart or lung disease. However, the normal exclusion criteria for MRI exams will still be adhered to:

  1. subjects with pacemakers, medical implants, aneurysm clips, or imbedded metal fragments will be excluded because of potential effects of the magnetic field
  2. women who are pregnant or who may be pregnant will be excluded because of the potential of a high level of RF power deposition on the fetus
  3. subjects who may experience claustrophobia will be excluded because of their inability to remain in the magnet for the time required to complete the exam

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 35 healthy volunteers (21 years or older) and 25 cardiac MRI patients of different age groups.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2006-08; Primary Completion 2010-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
cardiac motion reduction in cardiac MRI images | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: William Mahle, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States